CLINICAL TRIAL: NCT00520520
Title: Influence of Mild Therapeutic Hypothermia on Leukocyte Count
Acronym: INCA
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Charite University Medicine, Charite University Medicine
Other Study IDs: I-STU-26
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2009-07

CONDITIONS: Ventricular Fibrillation
Keywords: post resuscitation; post ventricular fibrillation; patients receiving mild therapeutic hypothermia
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Mild therapeutic hypothermia is indicated in patients surviving out-of-hospital cardiac arrest due to ventricular fibrillation. Potential immunologic responses are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of cardiac arrest due to VF
* Age 18-90

Exclusion Criteria:

* Suspected / proven pregnancy
* Immunodeficiency

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Survivors in out of hospital cardiac arrest
Sampling Method: Probability Sample
Dates: Start 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Schefold, MD, Principal Investigator — Charite University, Berlin, Germany; Christian Storm, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite University Hospital, Berlin, State of Berlin, Germany